CLINICAL TRIAL: NCT03972449
Title: The Impact of Beatboxing on the Management of Individuals With Residual Speech Errors
Brief Title: Beatboxing and Residual Speech Errors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not received.
Sponsor: Duquesne University (Other)
Responsible Party: Principal Investigator, Heather Leavy Rusiewicz, Associate Professor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DuquesneR21MusicHealth
Record Dates: First submitted 2019-02-27; First posted 2019-06-03 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Speech Sound Disorder
MeSH Terms: conditions — Speech Sound Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beatboxing: BEAT-Speech (Experimental)
  Interventions: Behavioral: BEAT-Speech
- Traditional Articulation Approach (Experimental)
  Interventions: Behavioral: Traditional Articulation Approach

INTERVENTIONS:
Behavioral: BEAT-Speech — BEAT-Speech integrates beatboxing techniques within speech-therapy services for individuals with speech sound disorders.
  Arms: Beatboxing: BEAT-Speech
Behavioral: Traditional Articulation Approach — The traditional approach to treating speech sound disorders focus on one or two sounds at a time until they are mastered by the client. Perceptual and production training are used with target starting at simple (isolation) and moving to more complex (sentences). A variety of cues such as shaping and phonetic placement cues are used.
  Arms: Traditional Articulation Approach

SUMMARY:
This project will study the effect of practicing speech sounds via beatboxing on speech accuracy, engagement in therapy, and functional outcomes for older children and adolescents with speech sound disorders (SSDs). Though SSDs exhibited by young children are often considered, SSDs are among the most frequent communication disorders in school-aged and adolescent children. SSDs can persist until adulthood. Individuals exhibit residual speech errors (RSE) when speech sounds are produced incorrectly after the age of eight, the age at which speech production is expected to be error-free. Common RSE include /r/, /s/, and /z/, all of which have high frequency in American English.

Beatboxing is a unique manipulation of the speech mechanism in which the individual creates repetitive, percussive and other instrumental sounds by actually being the instrument. Beatboxing is engaging and increasingly found in a variety of musical contexts and mainstream culture. The broad objective of this investigation is to explore the impact of beatboxing as an intervention tool on the speech produced and the functional outcomes attained by children with RSE compared to a traditional articulation therapy approach.The effect of a beatboxing intervention approach (BEAT-Speech) will be compared to traditional articulation therapy and employs a two-group pretest-posttest design. Specifically, the research aims to 1) assess the impact of beatboxing on speech sound production accuracy and amount of targets produced during therapy; 2) examine the relative level of client engagement of individuals exposed to beatboxing intervention; and 3) explore influences of beatboxing experiences on communication, activities, and participation in social and daily interactions.

ELIGIBILITY:
Inclusion Criteria:

• diagnosed with a speech sound disorder due to residual speech sound errors

Exclusion Criteria:

* out of age range
* history of hearing, neurogenic, behavioral diagnoses that can contribute to speech disorder
* English is not first or preferred language
* concurrent treatment for speech goals

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Speech sound accuracy: dichotomous ratings | within two years
  rated by naive, blinded raters
Speech sound accuracy: visual analog scale ratings | within two years
  rated by naive, blinded raters, will mark accuracy on a scale from 0-100 mm (not at all accurate to completely accurate). There is no formal name to this scale at this time given that it is novel to the study.
Phonetic accuracy | within two years
  % of consonants correct determined by phonetic transcription completed by trained transcribers

SECONDARY OUTCOMES:
therapeutic engagement level | within two years
  measured via clinician ratings and naive, blinded raters who will code nonverbal behaviors associated with engagement/disengagement
Hopkins Rehabilitation Engagement Rating | within two years
  five item quantitative questionnaire completed by instructors only after final session
Pittsburgh Rehabilitation Rating Scale | within two years
  single item questionnaire completed by instructors after each treatment session
PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Peer Relationship Scale | within two years
  questionnaire completed by participants to assess impact of treatment on social activities and participation. Scale is from 0-4 which is from worse to best outcome.
Adolescent Communication Questionnaire | within two years
  assesses self-efficacy/individual's belief in their ability to make change and succeed in therapy. Scale is fro 1 to 5 with the lowest number being associated with the greatest amount of negative impact to the highest number being associated with no impact.
Qualitative interview regarding functional outcomes | within two years
  phenomenological approach to better understanding themes associated with this novel therapy approach and traditional therapy approach

IPD SHARING:
Plan to Share IPD: No